CLINICAL TRIAL: NCT05749874
Title: Assess the Effects of Berberine on Preventing Cardiovascular Disease and Diabetes Mellitus Among Individuals With High Cardiometabolic Risk
Brief Title: Effects of Berberine on Preventing Cardiovascular Disease and Diabetes Mellitus
Acronym: ABCD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-CXGC04-1
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes; Abdominal Obesity; Hypertension; Dyslipidemias; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Prediabetic State; Obesity, Abdominal; Hypertension; Dyslipidemias; Atherosclerosis | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine group (Experimental): Berberine hydrochloride plus lifestyle intervention
  Interventions: Drug: Berberine plus lifestyle intervention
- placebo group (Placebo Comparator): Placebo plus lifestyle intervention
  Interventions: Behavioral: Placebo plus lifestyle intervention

INTERVENTIONS:
Drug: Berberine plus lifestyle intervention — berberine hydrochloride 500mg twice a day plus lifestyle intervention. Lifestyle intervention is based on Chinese guideline for primary prevention of cardiovascular diseases, and Chinese guideline for management of type 2 diabetes mellitus, coronary heart disease, myocardial infarction and stroke. Intervention includes health education on smoking, alcohol consumption, diet, physical activity and weight loss, etc.
  Arms: berberine group
Behavioral: Placebo plus lifestyle intervention — Placebo with identical shape, colour, odour and taste twice a day plus lifestyle intervention. Lifestyle intervention is based on Chinese guideline for primary prevention of cardiovascular diseases, and Chinese guideline for management of type 2 diabetes mellitus, coronary heart disease, myocardial infarction and stroke. Intervention includes health education on smoking, alcohol consumption, diet, physical activity and weight loss, etc.
  Arms: placebo group

SUMMARY:
This multicenter, double-blinded, randomized controlled trial aims to evaluate the effect of berberine on preventing cardiovascular disease and diabetes mellitus among individuals with high cardiometabolic risk in China.

DETAILED DESCRIPTION:
The trial aims to evaluate the efficacy and safety of berberine treatment for individuals with high cardiometabolic risk. Potential eligible patients will be recruited from about 100 medical centers in China. After a 4-to-6-week run-in period with berberine, all the eligible participants will be randomized (1:1) to berberine 500mg twice a day plus lifestyle intervention (Arm A) or placebo plus lifestyle intervention (Arm B). The participants will be followed up at month 3 and month 6, and once every 3 months thereafter, and be followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥40 years old
* Participants with prediabetes, defined as glycated hemoglobin (HbA1c) between 5.7% and 6.4%
* Participants with body mass index>25kg/m2, or abdominal obesity (i.e., waist circumference ≥85 cm in female or waist circumference ≥90 cm in male)
* Participants with established atherosclerosis cardiovascular diseases (ASCVD), or with at least two cardiovascular risk factors: (a) hypertension (b) aged ≥45(male) / 55 (female), (c) current smoker, (d) HDL-C<1mmol/L or TG≥2.3mmol/L
* Participants with established ASCVD required LDL-C≤70 mg/dL (1.8mmol/L) for participants with ASCVD or receiving optimized LDL-C-lowering therapy (at least moderate-intensity statin therapy, unless contraindicated or intolerant)

Exclusion Criteria:

* Participants with FPG≥7.0 mmol/L, diagnosed with diabetes or taking oral glucose-lowering drugs
* Participants diagnosed with acute coronary syndrome, stroke, transient ischemic attack, or undergoing cardiac surgery or cardiac intervention (i.e., implantation of cardiac closure devices, cardiac resynchronization therapy, or catheter ablation), percutaneous coronary intervention or valvuloplasty/other cardiac valve repair or implantation surgery within the 3 months before randomization
* Participants who plan to perform coronary and/or non coronary revascularization surgery, or cardiac surgery within 6 months after randomization
* Participants diagnosed with heart failure or left ventricular ejection fraction<40%, severe cardiac valvular disease, cardiomyopathy, congenital heart disease
* Conditions known to interfere with the accuracy of HbA1c measurement, including rheumatoid arthritis, hemolytic anemia, aplastic anemia, hemoglobinopathies, splenomegaly, splenectomy, vitamin B12 deficiency, alcoholism, long-term high-dose aspirin use, or chronic use of anesthetics or hydroxyurea
* Recipients of major organ transplants (e.g., lung, liver, heart, bone marrow, kidneys, etc.)
* Participants diagnosed with glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Participants taking berberine or drug containing berberine in the past 1 month
* Participants with any adverse reaction to berberine
* Participants with severe constipation, diarrhea, and/or severe chronic intestinal diseases (e.g., ulcerative colitis, Crohn's disease, irritable bowel syndrome, etc.)
* Participants who plan to have weight loss surgery, plan to take or currently taking drugs for weight loss
* Participants with active liver diseases, or alanine aminotransferase (ALT) / aspartate aminotransferase (AST) > 3 times upper limit of normal
* Estimated glomerular filtration rate (eGFR) < 45 ml/(min×1.73m2)
* Women who are pregnant or breastfeeding, or those who plan to be pregnant during the trial
* Participants with malignant tumors, or other serious diseases with life expectancy of less than 3 years
* Participants with mental disorders, cognitive disorders, or other serious diseases that could affect study participation
* Participants who participated or have been participating other trials during the last 3 months
* Any other conditions that may hinder the compliance to the study intervention or follow-up visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2024 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The distribution of glycemic status at 1 year after randomization | Intervention Period: 1 year
  Categorized as normal glucose metabolism, prediabetes, and diabetes

SECONDARY OUTCOMES:
Changes of glycemic-related parameters | Intervention Period: 1 year
  Including hemoglobin A1c (HbA1c), fasting plasma glucose (FPG), homeostasis model assessment of insulin resistance (HOMA-IR), and homeostasis model assessment of β-cell function (HOMA-β)
Changes of lipid-related parameters | Intervention Period: 1 year
  Including total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG), and lipoprotein(a)
Change of inflammation-related marker | Intervention Period: 1 year
  Including high-sensitivity C-reactive protein (hs-CRP)
Change of physical examination measures | Intervention Period: 1 year
  Including body mass index (BMI) and waist circumference
Changes of other parameters | Intervention Period: 1 year
  Including urinary albumin-to-creatinine ratio (UACR), serum uric acid, and metabolic syndrome score
Change of depressive symptoms | Intervention Period: 1 year
  Measured by Patient Health Questionnaire-9 (PHQ-9)
Time to first occurrence of composite endpoint of major cardiovascular event and diabetes | Intervention Period: 1 year
  cardiovascular death, non-hemorrhagic stroke, myocardial infarction, arterial revascularization, and diabetes
Time to new-onset diabetes | Intervention Period: 1 year
  Diabetes is determined by oral glucose tolerance test, clinical diagnosis or use of glucose-lowering medications.
Normalization of glucose parameters | Intervention Period: 1 year
  Meeting all three criteria: 1) Fasting plasma glucose (FPG)<6.1 mmol/L; 2) 2-hour postprandial blood glucose (2hPG)<7.8 mmol/L; 3) HbA1c<5.7%.
Time to newly diagnosed cancer | Intervention Period: 1 year
  all events of cancer or classified by primary sites
Exploratory biomarker analyses | Intervention Period: 1 year
  Including serum trimethylamine, trimethylamine N-oxide, dopamine, berberine metabolites, and lipidomics analyses; urinary berberine metabolite analyses; and gut microbiota sequencing analyses.
Time to first occurrence of composite endpoint of major cardiovascular event and diabetes | Entire follow-up period: 4 years
  cardiovascular death, non-hemorrhagic stroke, myocardial infarction, arterial revascularization, and diabetes
Time to new-onset diabetes | Entire follow-up period: 4 years
  Diabetes is determined by oral glucose tolerance test, clinical diagnosis or use of glucose-lowering medications.
Time to first occurrence of composite endpoint of major cardiovascular event 1 | Entire follow-up period: 4 years
  cardiovascular death, non-hemorrhagic stroke, myocardial infarction, arterial revascularization
Time to first occurrence of composite endpoint of major cardiovascular event 2 | Entire follow-up period: 4 years
  cardiovascular death, non-hemorrhagic stroke, myocardial infarction
Time to newly diagnosed cancer | Entire follow-up period: 4 years
  all events of cancer or classified by primary sites

OTHER OUTCOMES:
Subgroup analysis 1 for primary outcome measure | Intervention Period: 1 year
  Age (<55，55-65，≥65)
Subgroup analysis 2 for primary outcome measure | Intervention Period: 1 year
  Sex (male, female)
Subgroup analysis 3 for primary outcome measure | Intervention Period: 1 year
  Body mass index (<28kg/m2, ≥28kg/m2)
Subgroup analysis 4 for primary outcome measure | Intervention Period: 1 year
  Statin use (yes, no)
Subgroup analysis 5 for primary outcome measure | Intervention Period: 1 year
  HbA1c median
Subgroup analysis 6 for primary outcome measure | Intervention Period: 1 year
  Hs-CRP tertiles
Subgroup analysis 7 for primary outcome measure | Intervention Period: 1 year
  LDL-C tertiles
Subgroup analysis 8 for primary outcome measure | Intervention Period: 1 year
  Triglyceride tertiles
Subgroup analysis 9 for primary outcome measure | Intervention Period: 1 year
  HDL-C tertiles
Safety assessment during the intervention period | Intervention Period: 1 year
  Including serious adverse events, non-serious adverse events of special interest, and treatment discontinuation for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Haibo Zhang, MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, National Center for Cardiovascular Diseases, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
All the IPD that underlie results in the publication with study protocol and SAP will be shared to the public on the study website upon request with a protocol after approval from the ABCD steering committee. The access criteria and URL of the study website is not established yet.

REFERENCES:
- [Background] Kong WJ, Vernieri C, Foiani M, Jiang JD. Berberine in the treatment of metabolism-related chronic diseases: A drug cloud (dCloud) effect to target multifactorial disorders. Pharmacol Ther. 2020 May;209:107496. doi: 10.1016/j.pharmthera.2020.107496. Epub 2020 Jan 27. PMID 32001311
- [Background] Kong W, Wei J, Abidi P, Lin M, Inaba S, Li C, Wang Y, Wang Z, Si S, Pan H, Wang S, Wu J, Wang Y, Li Z, Liu J, Jiang JD. Berberine is a novel cholesterol-lowering drug working through a unique mechanism distinct from statins. Nat Med. 2004 Dec;10(12):1344-51. doi: 10.1038/nm1135. Epub 2004 Nov 7. PMID 15531889